CLINICAL TRIAL: NCT00499642
Title: A Single-Dose, Double-Blind, Crossover, Placebo- and Moxifloxacin (Open-Label)-Controlled Study of the Effects of Lecozotan SR on Cardiac Repolarization in Healthy Adult Subjects
Brief Title: Study Evaluating the Effect of Lecozotan SR on the QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3098B1-133
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer Disease; Healthy
Keywords: Healthy Subjects
MeSH Terms: conditions — Alzheimer Disease | interventions — lecozotan; Moxifloxacin

INTERVENTIONS:
Drug: Lecozotan SR
Drug: Moxifloxacin

SUMMARY:
This is a randomized, double-blind, placebo- and moxifloxacin (open-label)-controlled, 4-period crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18 to 55 years inclusive.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of any clinically important drug allergy.
* Positive findings of urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-06; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To assess the effect of drug administration on QTc interval.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France: infomedfrance@wyeth.com
Locations (2):
- France (2):
  - Rennes
  - Rueil-Malmaison